CLINICAL TRIAL: NCT07160920
Title: A Risk Score for Prediction of Gestational Diabetesmellitus in China Using Routinely Collected Hospital Data
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-2763
Record Dates: First submitted 2025-07-03; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes Mellitus (GDM)
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant woman
  Interventions: Other: Collect clinical data of pregnant women

INTERVENTIONS:
Other: Collect clinical data of pregnant women — Collect clinical data of pregnant women

SUMMARY:
This project will recruit 6,608 pregnant women in the early stage of pregnancy in Beijing and across the country. Researchers (prenatal examination doctors) will collect the basic information of pregnant women and the results of early pregnancy laboratory tests through hospital systems (HIS and LIS systems). The dietary frequency and exercise information of pregnant women were collected through questionnaire surveys: A 75g oral glucose tolerance test (0GTT test) was conducted at 24-28 weeks. Follow-up was conducted until the completion of the 75gOGTT test, and the delivery outcomes were recorded. By making the subjects pay attention to their own physical conditions through the project, abnormalities can be detected early. At the same time, early prediction of gestational diabetes mellitus enables doctors and health physicians to identify high-risk groups for gestational diabetes mellitus (GDM) at an early stage and carry out early intervention, reducing GDM and related pregnancy complications, promoting the health of mothers and infants, and reducing the additional medical expenses that may be borne for GDM management and the overall medical expenditure of the country in the future.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with single pregnancies in the early stage of pregnancy who have registered in the hospital are eligible to participate in the proposed program.

Exclusion Criteria:

Pregnant women with a known history of type 1 or type 2 diabetes will be excluded.

Ages: 21 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: All pregnant women who have registered their medical records at Peking Union Medical College Hospital and have not had diabetes before pregnancy are eligible to participate in this project
Sampling Method: Probability Sample
Enrollment: 6608 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Complications during pregnancy | During childbirth
mode of delivery | During childbirth
premature rupture of membranes | During childbirth
The length of a newborn | During childbirth
Newborn weight | During childbirth
apgar score | During childbirth

OTHER OUTCOMES:
Ultrasound examination results such as fetal biparietal diameter, head circumference, abdominal circumference and femoral length (unit: mm). | From 28 weeks of gestation until delivery
Clinical Laboratory Indicators | 4 to 7 weeks of gestation, 24 to 28 weeks of gestation, and 37 to 38 weeks of gestation
height of pregnant women | Baseline
weight of pregnant women | Baseline
BMI of pregnant women | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No